CLINICAL TRIAL: NCT01739309
Title: Phase 2 Study of a CDK4/6 Inhibitor for Patients With Relapsed or Refractory Mantle Cell Lymphoma
Brief Title: Study of LY2835219 for Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13269; I3Y-MC-JPBB (Other: Eli Lilly and Company); 2012-003614-14 (EudraCT Number)
Record Dates: First submitted 2012-11-29; First posted 2012-12-03 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Mantle Cell Lymphoma
Keywords: Non- Hodgkins Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin | interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abemaciclib (Experimental): 200 milligram (mg) abemaciclib administered orally every 12 hours on days 1 through 28 of a 28-day cycle
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — Administered orally
  Other Names: LY2835219

SUMMARY:
The purpose of this study is to estimate the disease control rate with abemaciclib for relapsed or refractory mantle cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of relapsed or refractory Mantle Cell Lymphoma (MCL) according to the World Health Organization (WHO) classification that has relapsed after, or been refractory to, available standard treatments. However, participants who are intolerant of, or unable to receive a standard treatment are not required to have MCL that has relapsed after, or been refractory to, that specific standard treatment. Pathology must be reviewed and confirmed at the investigational site where participant is entered prior to enrollment
* Have disease that is assessable according to the Response Criteria for Non- Hodgkin's Lymphomas
* Have given written informed consent prior to any study-specific procedures
* Have adequate organ function including:

  * Hematologic: Absolute neutrophil count (ANC) ≥1.5 x 10^9/Liter (L), platelets ≥75 x 10^9/L, and hemoglobin ≥8 grams per deciliter (g/dL)
  * Hepatic: Bilirubin ≤1.5 times upper limits of normal (ULN) and alanine aminotransferase (ALT) ≤3.0 times ULN
  * Renal: Estimated creatinine clearance ≥50 milliliter per minute (ml/min)
* Have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1, or 2
* Have discontinued all previous therapies for cancer (including chemotherapy, radiotherapy, immunotherapy, and investigational therapy) for at least 21 days for myelosuppressive agents or 14 days for nonmyelosuppressive agents prior to receiving study drug, and recovered from the acute effects of therapy (treatment-related toxicity resolved to baseline) except for residual alopecia
* Are willing to make themselves available for the duration of the study and to follow study procedures
* Are amenable to compliance with protocol schedules and testing
* Males and females with reproductive potential must agree to use medically approved contraceptive precautions during the trial and for 3 months following the last dose of study drug
* Females with child-bearing potential must have a negative serum pregnancy test within 14 days of the first dose of study drug
* Have a life expectancy of ≥12 weeks
* Are able to swallow capsules

Exclusion Criteria:

* Are currently enrolled in, or discontinued within 14 or 21 days of the initial dose of study drug for a nonmyelosuppressive or myelosuppressive agent, respectively, a clinical trial involving an investigational product or non-approved use of a drug or device other than the study drug used in this study, or concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study
* Have serious preexisting medical conditions that, in the judgment of the investigator, would preclude participation in this study (for example, pneumonia, inflammatory bowel disease, history of major surgical resection involving the stomach or small bowel)
* Have symptomatic metastasis to the central nervous system (CNS). Participants may have CNS metastasis that is radiographically or clinically stable for at least 14 days prior to receiving study drug, regardless of whether they are receiving corticosteroids
* Have received an autologous or allogeneic stem-cell transplant within 75 days of the initial dose of study drug. In addition, recipients of an allogenic stemcell transplant must have discontinued immunosuppressive therapy at least 14 days before study drug administration with no more than Grade 1 acute graft versus-host disease on Day 1 of Cycle 1
* Females who are pregnant or lactating
* Have active bacterial, fungal, and/or known viral infection (for example, human immunodeficiency virus [HIV] antibodies, hepatitis B surface antigen [HBSAg], or hepatitis C antibodies). Screening is not required for enrollment
* Have a baseline electrocardiogram (ECG) with any of the following findings: ventricular tachycardia, ventricular fibrillation, abnormal QTcB (defined as ≥450 milliseconds for males and ≥470 milliseconds for females), or evidence of acute myocardial ischemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-03-20 (Actual); Primary Completion 2015-09-28 (Actual); Study Completion 2022-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- France (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pessac
- Germany (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Homburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kassel
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mainz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nuremberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ulm

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Gelbert LM, Cai S, Lin X, Sanchez-Martinez C, Del Prado M, Lallena MJ, Torres R, Ajamie RT, Wishart GN, Flack RS, Neubauer BL, Young J, Chan EM, Iversen P, Cronier D, Kreklau E, de Dios A. Preclinical characterization of the CDK4/6 inhibitor LY2835219: in-vivo cell cycle-dependent/independent anti-tumor activities alone/in combination with gemcitabine. Invest New Drugs. 2014 Oct;32(5):825-37. doi: 10.1007/s10637-014-0120-7. Epub 2014 Jun 13. PMID 24919854

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers are those who died, or are alive and being followed at the end of the trial but off treatment.
Groups:
- Abemaciclib: 200 milligram (mg) of Abemaciclib was administered orally every 12 hours on days 1 through 28 of a 28-day cycle
Period: Overall Study
Arm/Group | Abemaciclib
Started | 28
Received at Least One Dose of Study Drug | 28
Completed | 26
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Abemaciclib: 200 mg Abemaciclib was administered orally every 12 hours on days 1 through 28 of a 28-day cycle
Arm/Group | Abemaciclib
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 28
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 27
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  France | 13
  Germany | 15

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieve Disease Control Rate (DCR) Which Includes Complete Response (CR), Complete Response Unconfirmed (CRu), Partial Response (PR) or Stable Disease (SD)
Description: The DCR was estimated based on the Response Criteria for Non-Hodgkin's Lymphomas (Cheson et al. 1999). DCR was assessed from date of first dose until disease progression or death or start of new anticancer therapy. CR is defined as the disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms based on CT scan or bone marrow biopsy; CRu = the CR criteria is met and a residual lymph node mass greater than 1.5 cm in greatest transverse diameter that has regressed by more than 75% in the sum of the product diameter (SPD). PR is >= 50% decrease in SPD of the six largest nodal masses/no new sites of disease. Progressive Disease (PD) is defined as an increase by 25% in longest diameter, new lesion or assessable disease progression. SD=small changes not meeting the above criteria; DCR and its exact 95% confidence interval (CI) was estimated for treated participants using the Clopper-Pearson method.
Time Frame: From Date of First Dose until Disease Progression or Death or Start of New Anticancer Therapy (Up to 28 Months)
Population: All participants who received at least one dose of study drug and had evaluable DCR data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abemaciclib
Number analyzed (Participants) | 28
percentage of participants | 71.4 [51.3 to 86.8]

2. Secondary Outcome: Percentage of Participants Who Achieve Best Overall Disease Response (BOR) That Includes CR, CRu or PR
Description: BOR was assessed based on the Response Criteria for Non-Hodgkin's Lymphomas and was measured from date of first dose until the earliest evidence of objective progression or start of new anticancer therapy. Any responses observed after objective progression or after the start of new anticancer therapy are excluded from the determination of best response. A second confirmatory radiological tumor assessment was performed at least 28 days after the first evidence of response (CR, CRu, or PR). Two objective status determinations of CR (or CRu) before progression were required for a best response of CR (or CRu). Two determinations of PR or better before progression, but not qualifying for CR or CRu, were required for a best response of PR.
Time Frame: From Date of First Dose until Disease Progression (Up to 28 Months)
Population: All participants who received at least one dose of study drug and had evaluable BOR data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Abemaciclib
Number analyzed (Participants) | 28
percentage of participants | 35.7 [18.6 to 55.9]

3. Secondary Outcome: Duration of Objective Response (DOR)
Description: DOR is from the date when criteria for objective response (ie, CR, CRu or PR) are met, to the first documentation of relapse or disease progression or death due to any cause. DOR is based on the Response Criteria for Non-Hodgkin's Lymphomas of the Cancer and Leukemia Group B. CR is defined as disappearance of all disease, no symptoms and must last 4 weeks or "unconfirmed CR, (CRu)". PR is defined as >= 50% decrease in sum of product diameter (SPD), no increase or new lesion, or assessable disease stable or decreased, must last 4 weeks or CRu. Progressive Disease or PD is defined as an increase by 25% in longest diameter, new lesion, or assessable disease progression. DOR was analyzed using Kaplan-Meier methods. If the participant receives other anticancer therapy prior to progression, the participant was censored at the start date of this other therapy.
Time Frame: From Date of CR, CRu or PR until Disease Progression or Death Due to Any Cause (Up to 28 Months)
Population: All participants who received at least one dose of study drug and achieved BOR. 4 participants were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abemaciclib
Number analyzed (Participants) | 10
months | 12.39 [3.19 to NA] — The upper limit of the 95% CI was not calculated due to the high censoring rate.

4. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the date of first dose until disease progression or death due to any cause based on the Response Criteria for Non-Hodgkin's Lymphomas. Disease progression is defined as the first date of documentation of a new lesion or enlargement of a previous lesion, or the date after radiologic assessment has been completed. PD is defined as an increase by 25% in longest diameter, new lesion, or assessable disease progression. Progression-free survival was analyzed using Kaplan-Meier methods. If the participant receives other anticancer therapy prior to progression, the participant was censored at the start date of this other therapy.
Time Frame: From Date of First Dose until Disease Progression or Death Due to Any Cause (Up to 28 Months)
Population: All participants who received at least one dose of study drug. 9 participants were censored.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib
Number analyzed (Participants) | 28
Months | 8.18 [4.34 to 16.03]

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as from the date of first dose until death due to any cause. For each participant who is not known to have died as of the data-inclusion cutoff date for overall survival analysis, OS were censored on the last date the participant is known to be alive. Overall survival was analyzed using Kaplan-Meier methods.
Time Frame: From Date of First Dose until Death Due to Any Cause (Up to 28 Months)
Population: All participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib
Number analyzed (Participants) | 28
Months | 16.03 [6.77 to NA] — The 95% confidence interval upper limit was not reached (NR).

6. Secondary Outcome: Event-Free Survival
Description: Event-free survival (time to treatment failure) is measured from date of first dose to disease progression, or discontinuation of treatment for any reason (eg, disease progression, toxicity, participant preference, initiation of new treatment without documented progression, or death due to any cause). 2 participants were censored. Event-free survival is defined only for responders (participants with a CR, CRu, or PR).
Time Frame: From Date of First Dose until Disease Progression, Discontinuation of Treatment, or Death Due to Any Cause (Up to 28 Months)
Population: All participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Abemaciclib: 200 mg was Abemaciclib administered orally every 12 hours on days 1 through 28 of a 28-day cycle.
Arm/Group | Abemaciclib
Number analyzed (Participants) | 28
Months | 11.29 [5.45 to 16.26]

7. Secondary Outcome: Time to Disease Progression
Description: Time to Disease Progression is based on the response criteria of Non-Hodgkin's Lymphomas. Time to progression (TTP) is defined as the time from date of first dose until documented disease progression or death as a result of lymphoma. In TTP, deaths from other causes are censored either at the time of death or at an earlier time of assessment.
Time Frame: From Date of First Dose Until Disease Progression (Up to 28 Months)
Population: All participants who received at least one dose of study drug. 17 participants were censored.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib
Number analyzed (Participants) | 28
Months | 12.85 [5.45 to NA] — The upper limit was not calculated due to the high censoring rate.

8. Secondary Outcome: Disease-Free Survival
Description: Disease-free survival is measured from first dose until date of disease progression or the time of occurrence of disease-free state or attainment of a CR to disease recurrence or death as a result of lymphoma or acute toxicity of treatment. Progressive Disease (PD) is defined as an increase by 25%, new lesion, or accessible progressive disease. Disease-Free Survival was assessed based on the response criteria of Non-Hodgkins Lymphomas. Disease-free survival is only defined for participants with response.
Time Frame: First Dose Until Date of Disease Progression or Time of Occurrence Disease-Free State or CR to Disease Recurrence or Death (Up to 28 Months)
Population: All participants who received at least one dose of study drug. 5 participants were censored.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abemaciclib
Number analyzed (Participants) | 28
Months | 9.20 [3.19 to NA] — The 95% confidence interval upper limit was not reached (NR).

9. Secondary Outcome: Change From Baseline in Functional Assessment of Cancer Therapy - Lymphoma (FACT-Lym) TOI and Subscale Scores
Description: Change From Baseline in FACT-Lym Total Outcome Index (TOI) Score (Follicular Lymphoma Population). The FACT-Lym TOI Score for the follicular lymphoma population was derived from the following 3 individual FACT-Lym questionnaire subscale scores: Physical Well-being (range: 0-28), Functional Well-being (range: 0-28) and Lymphoma (range: 0-60). The FACT-Lym TOI Score is the sum of the 3 individual subscales (range 0-116). Higher scores indicate better outcomes and lower scores indicate worse outcomes. A positive change from baseline indicates an improvement and a negative change is a detriment.
Time Frame: Baseline, Cycle 5 (Up To Day 140)
Population: All participants who received at least one dose of study drug and had baseline and post baseline FACT-Lym data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Abemaciclib
Number analyzed (Participants) | 13
units on a scale
  Physical Well-Being (PWB) Subscale Score | 0.2 (5.6)
  Functional (FWB) Subscale Score | -0.9 (4.5)
  LYM Subscale Score | 1.1 (5.2)
  FACT-Lym TOI Score | 0.5 (12.5)

10. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration (Cmax) of Abemaciclib
Time Frame: Predose, 1 hour (hr), 2 hr, 4 hr, 6 hr, 8 hr, 10 Hours Postdose
Population: All participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/ml)
Arm/Group | Abemaciclib
Number analyzed (Participants) | 26
nanogram/milliliter (ng/ml) | 189 (59)

11. Secondary Outcome: PK - Area Under the Concentration-Time Curve From Zero to Last Time Point (AUC[0-tlast]) of Abemaciclib
Time Frame: Predose, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 10 Hours Postdose
Population: All randomized who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanogram/milliliter (hr*ng/ml)
Arm/Group | Abemaciclib
Number analyzed (Participants) | 26
hour*nanogram/milliliter (hr*ng/ml) | 978 (61)

12. Secondary Outcome: PK - Terminal Half Life (T 1/2) of Abemaciclib
Time Frame: Predose, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 10 Hours Postdose
Population: Zero participants were analyzed due to the calculation of half-life (t1/2) by noncompartmental analysis was not possible due to cessation of sampling at 8 hours postdose.
Arm/Group | Abemaciclib
Number analyzed (Participants) | 0

13. Secondary Outcome: PK: Volume of Distribution (Vd) of Abemaciclib
Time Frame: Predose, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 10 Hours Postdose
Population: Zero participants were analyzed. Vd was not calculated by non-compartmental analysis with the available data.
Arm/Group | Abemaciclib
Number analyzed (Participants) | 0

14. Secondary Outcome: PK: Clearance (CL) of Abemaciclib
Time Frame: Predose, 1 hr, 2 hr, 4 hr, 6 hr, 8 hr, 10 Hours Postdose
Population: Zero participants were analyzed. CL was not calculated due to PK sampling schedule was not suitable for estimation of these PK parameters.
Arm/Group | Abemaciclib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Baseline till end of follow-up (Up to 7.9 years)
Description: All participants who received at least one dose of study drug.
Arm/Group | Abemaciclib
All-Cause Mortality (participants affected / at risk) | 23/28
Serious Adverse Events (participants affected / at risk) | 13/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib (N=28)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Ileus (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
General physical health deterioration (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (2)
Device related infection (Infections and infestations) | 1 (1)
Meningitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (3)
Progressive multifocal leukoencephalopathy (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nervous system disorder (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Abemaciclib (N=28)
Anaemia (Blood and lymphatic system disorders) | 8 (8)
Leukopenia (Blood and lymphatic system disorders) | 3 (5)
Neutropenia (Blood and lymphatic system disorders) | 7 (8)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (12)
Abdominal pain (Gastrointestinal disorders) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 21 (31)
Nausea (Gastrointestinal disorders) | 9 (14)
Vomiting (Gastrointestinal disorders) | 8 (56)
Asthenia (General disorders) | 2 (3)
Fatigue (General disorders) | 10 (15)
Oedema peripheral (General disorders) | 6 (8)
Pyrexia (General disorders) | 4 (5)
Bronchitis (Infections and infestations) | 6 (6)
Conjunctivitis (Infections and infestations) | 4 (4)
Nasopharyngitis (Infections and infestations) | 2 (4)
Rhinitis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 4 (6)
Blood creatinine increased (Investigations) | 7 (9)
Gamma-glutamyltransferase increased (Investigations) | 2 (9)
Neutrophil count decreased (Investigations) | 4 (12)
Platelet count decreased (Investigations) | 3 (4)
Weight decreased (Investigations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 4 (4)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2)
Dizziness (Nervous system disorders) | 4 (4)
Dysgeusia (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (3)
Presyncope (Nervous system disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days